CLINICAL TRIAL: NCT04071301
Title: An Explorative, Open, Single-arm Clinical Investigation to Collect Real-life Measurement Data in Order to Assess the Mathematical Algorithms Involved in TENA SmartCare Change Indicator.
Brief Title: Collection of Real-life Measurement Data for TENA SmartCare Change Indicator in Subjects With Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essity Hygiene and Health AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: FUEL_CIP_Ver.B_19-Jul-2019
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Results first posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational Device (Experimental): TENA SmartCare Change Indicator
  Interventions: Device: TENA SmartCare Change Indicator

INTERVENTIONS:
Device: TENA SmartCare Change Indicator — Each participating subject will be provided with a Change Indicator and absorbent products for the duration of the investigation. Nine types of absorbent products will be used to collect real-life measurement data in order to assess the mathematical algorithms involved in the TENA SmartCare Change Indicator. Each participating subject will be allocated to the type(s) that are considered most suitable.
  Gateways will be placed in the resident's rooms as well as in common areas, this to enable full measurement registration.

SUMMARY:
This study is an explorative, open, single-arm clinical investigation to collect real-life measurement data in order to assess the mathematical algorithms involved in TENA SmartCare Change Indicator.

DETAILED DESCRIPTION:
The purpose of this exploratory clinical investigation is to evaluate safety and to collect real-life measurement data using the TENA SmartCare Change Indicator. The collected data will be used to assess the device related algorithms. These algorithms have been established and verified in a laboratory environment. However, due to possible differences in parameters, real-life measurement data are to be collected to aid in further product development.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is willing and able to provide informed consent and to participate in the clinical investigation.
2. The subject is ≥18 years of age.
3. The subject is diagnosed with urinary incontinence.
4. The subject is being cared for at Tre Stiftelser.

Exclusion Criteria:

1. The subject has ≥ 4 fecal "incidences" per week.
2. The subject has severe absorbent product related skin problems, as judged by the investigator.
3. The subject is hyper sensitive related to allergic reaction to any of the included materials, as judged by the investigator.
4. The subject has ≥ 2 intermittent urinary catheters per day.
5. The subject has a pacemaker or an implantable cardioverter-defibrillator.
6. The subject removes the incontinence product.
7. The subject demonstrates responsive behavior towards sensors.
8. The subject has any other condition that may make participation in the clinical investigation inappropriate, as judged by investigator.
9. The subject is not cared for at Tre Stiftelser.
10. The subject is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Molander, MD, PhD, Principal Investigator — Avd. för Invärtes medicin och klinisk nutrition, Högsbo sjukhus, Göteborg
Locations (1):
- Tre Stiftelser, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled to the investigation on 05 September 2019. The last subject´s last visit was on 27 November 2019.The study was carried out at a nursing home.
Groups:
- Investigational Device: TENA SmartCare Urine Sensor and Gateway
  Each participating subject was provided with Urine Sensor and absorbent products for the duration of the investigation. Seven types of absorbent products were used to collect real-life measurement data in order to assess the mathematical algorithms involved in the TENA SmartCare Change Indicator. Each participating subject was allocated to the type(s) that were considered most suitable.
  Gateways were placed in the resident's rooms as well as in common areas to enable full measurement registration.
Period: Overall Study
Arm/Group | Investigational Device
Started | 15
Completed | 8
Not Completed | 7
Not completed — Withdrawal by Subject | 6
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set Population (FAS). Of the 15 subjects enrolled and found to be eligible for participation, incontinence products registrations were obtained from 13 subjects and thereby included in the FAS.
Groups:
- Investigational Device: TENA SmartCare Urine Sensor and Gateway
Arm/Group | Investigational Device
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 84 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 13
Bedridden [Count of Participants; unit: Participants] | 1
Childbearing potential of subjects [Count of Participants; unit: Participants] | 0
Number of subjects with general health status assessed as fair [Count of Participants; unit: Participants] — Poor, fair, good, very good.
  Participants | 13
Prior use of incontinence products [Count of Participants; unit: Participants] — Number of subjects that used incontinence products developed by Essity 6 months prior to baseline.
  Participants | 1

OUTCOME MEASURES:

1. Primary Outcome: Urine Volume Quantification and Impedance Measurements
Description: Descriptive statistics were used to summarize any individual differences between the predicted urine volume from the Change Indicator and the true urine volume (by measuring absorbent product weight). A measure of mean difference for the predicted volume minus true volume is assessed. A combination of these values were used to assess the mathematical algorithms for the TENA SmartCare Change Indicator.
Time Frame: 11 weeks
Population: Full Analysis Set (FAS) include data from 13 out of 15 subjects. 684 out of 1180 collected data points were included in the primary endpoint analysis.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Investigational Device
Number analyzed (Participants) | 13
ml | 46 (213)

ADVERSE EVENTS:
Time Frame: 11 weeks
Groups:
- Investigational Device: TENA SmartCare Urine Sensor and Gateway
  .
Arm/Group | Investigational Device
All-Cause Mortality (participants affected / at risk) | 1/15
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Device (N=15)
Choke (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stroke (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Only the Change indicator and Gateway were used, i.e. the smart phone app was not part of the investigation why the clinical benefit relating to app notifications was not investigated. There was a drop off in eligible data points compared to the total number of data points. The reason to this was device deficiencies on some sensors leading to erroneous raw data. The deficiencies were anticipated as the sensors being pre-production devices. 2/3 of the data points were used for evaluation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT04071301/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-27): https://cdn.clinicaltrials.gov/large-docs/01/NCT04071301/SAP_001.pdf